CLINICAL TRIAL: NCT04131179
Title: Youth Culturally Adapted Manual Assisted Psychological Therapy (Y-CMAP) in Adolescents Pakistani Patients With a History of Self Harm
Brief Title: Multicenter Study to Evaluate the Clinical and Cost Effectiveness of a Youth Culturally Adapted Therapy (YCMAP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Collaborators: University of Manchester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PILL-YCMAP-001
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Self Harm
Keywords: Self-harm, adolescents, adaptation, problem solving, LMICs
MeSH Terms: conditions — Self-Injurious Behavior | interventions — Psychosocial Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Youth culturally adapted therapy (Y-CMAP) (Experimental): Youth Culturally adapted manual assisted (Y-CMAP) psychological therapy
  Interventions: Behavioral: Youth Culturally Adapted Manual Assisted Psychological Therapy (Y-CMAP)
- Treatment as Usual (No Intervention): TAU will be standard routine care delivered by local medical, psychiatric and primary care services according to clinical judgement. A record will be kept of any treatment received by each participant.
  Assessment will be done at 3rd,6th,9th and 12 month after randomization along with TAU

INTERVENTIONS:
Behavioral: Youth Culturally Adapted Manual Assisted Psychological Therapy (Y-CMAP) — Y-CMAP is a manual assisted brief psychological intervention based on the principles of Cognitive Behaviour Therapy (CBT), including 8-10 sessions delivered over three months.
  This intervention includes evaluation of the self-harm attempt, psycho education, crisis skills, problem solving and simple cognitive techniques to manage emotions, negative thinking,relapse prevention strategies and training on anger management and assertiveness.
  Other Names: Psychosocial Intervention
  Arms: Youth culturally adapted therapy (Y-CMAP)

SUMMARY:
To evaluate the clinical and cost-effectiveness of a youth culturally adapted manual assisted therapy (YCMAP) in Pakistani Adolescents with a history of self-harm

DETAILED DESCRIPTION:
Globally suicide is the second leading cause of death in young people 15-29 years of age. A recent review indicated that the reported suicide rates in South Asia are high compared to the global average. These figures are likely to be an under estimate since suicide data from many Low and Middle Income Countries (LMICs) is lacking. There is little official data on suicide from Pakistan, where suicide and self-harm remains as criminal act and socially, religiously condemned. However, there is accumulating evidence that both self-harm and suicide rates have been increasing in Pakistan.

This is the first RCT of a psychological intervention for self-harm in children and young people in Pakistan. It follows from the work of "Multicentre RCT to evaluate the clinical and cost effectiveness of culturally adapted manual assisted psychological intervention"(CMAP) trial currently taking place in adults who have self-harmed in Pakistan, by evaluating whether a similar intervention, adapted for children and adolescents, could be clinically and cost effective.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 12-18 years presenting to the participating GPs, emergency departments or admitted after an episode of self-harm to the participating hospitals or self-referrals.
* History of recent self-harm. Recent self-harm is defined as self-harm occurring within the last 3 months (from the initial identification of a potential participant).
* Participants living within the catchment area of the participating practices and hospitals.
* Not needing inpatient psychiatric treatment.

Exclusion Criteria:

* Severe mental illness (such as Psychotic disorder) as Self-harm commonly co- occurs with other mental health difficulties.
* Conditions limiting engagement with assessment or intervention, including developmental and communication disorders, intellectual disabilities and autistic spectrum disorders.
* Temporary resident unlikely to be available for follow up.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 684 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2022-09-08 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Suicide Attempt Self Injury Interview SASII | Change in scores from baseline to 12th months
  Repetition rate of self-harm measured by adapted Suicide Attempt Self-Injury Interview (SASII). Higher number on repetition indicates worse outcome and vice versa

SECONDARY OUTCOMES:
Beck Scale for Suicidal ideation (BSI) | Change in scores from Baseline to 3rd, 6th, 9th and 12th month.
  Suicidal ideation will be assessed with the Beck Scale for Suicide Ideation (BSS; Beck & Steer, 1991), a 19-item self-report questionnaire, measuring the intensity and frequency of suicidal thoughts within the past week. Minimum total score is 0 and maximum total score can be 38. Higher scores indicate worse outcome.
Beck Hopelessness Scale | [Time Frame: Baseline,3rd,6th,9th and 12th months]
  This is a 20 items scale measuring hopelessness. Higher scores on the scale indicate greater severity of hopelessness. Minimum total score on this scale can be 0 and maximum total score can be 20, with higher levels of hopelessness indicated by higher scores on the scale.
Psychological Distress Scale | Change in scores from Baseline to 3rd, 6th, 9th and 12th month.
  It's a 10 item scale measuring emotional states with a 5 level response scale. The maximum score is 50 indicating severe distress, and the minimum score is 10 indicating no distress.
EuroQol-5 Dimensions (EQ5-D) | Change in scores from Baseline to 3rd, 6th, 9th and 12th month.
  A standardised instrument to measure health status and associated population utility weights. It consists of a self-report questionnaire covering five dimensions of health (mobility, self-care, usual activities, pain/ discomfort and anxiety/ depression).
Client Satisfaction Questionnaire (CSQ). | Change in scores from Baseline to 3rd, 6th, 9th and 12th month.
  The participants will rate their satisfaction with treatment by using the CSQ. The total score ranges from 8 to 32. Higher scores indicate higher level of satisfaction.
Client Services Receipt Inventory CSRI | Change in scores from Baseline to 3rd, 6th, 9th and 12th month.
  We will collect information on the use of health services (including the informal sector such as faith healers/Imams)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Nusrat Husain, MD, Principal Investigator — University of Manchester (OTHER SPONSOR_RESPONSIBLE PARTY)
Locations (3):
- Pakistan (3):
  - Karachi Site, Karachi, Sindh
  - Lahore Site, Lahore
  - Rawalpindi Site, Rawalpindi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Linehan MM, Comtois KA, Brown MZ, Heard HL, Wagner A. Suicide Attempt Self-Injury Interview (SASII): development, reliability, and validity of a scale to assess suicide attempts and intentional self-injury. Psychol Assess. 2006 Sep;18(3):303-12. doi: 10.1037/1040-3590.18.3.303. PMID 16953733
- [Background] Beck, A. T., & Steer, R. A. (1991). BSI, Beck scale for suicide ideation: manual: Psychological Corporation.
- [Background] Beck, A., & Steer, R. J. S. A., TX: Psychological Corporation. (1988). Manual for the Beck hopelessness scale
- [Background] Brooks R. EuroQol: the current state of play. Health Policy. 1996 Jul;37(1):53-72. doi: 10.1016/0168-8510(96)00822-6. PMID 10158943
- [Background] Andrews G, Slade T. Interpreting scores on the Kessler Psychological Distress Scale (K10). Aust N Z J Public Health. 2001 Dec;25(6):494-7. doi: 10.1111/j.1467-842x.2001.tb00310.x. PMID 11824981
- [Background] Attkisson CC, Zwick R. The client satisfaction questionnaire. Psychometric properties and correlations with service utilization and psychotherapy outcome. Eval Program Plann. 1982;5(3):233-7. doi: 10.1016/0149-7189(82)90074-x. PMID 10259963
- [Background] Beecham, J., & Knapp, M. J. M. m. h. n. (2001). Costing psychiatric interventions. 2, 200-224.
- [Derived] Husain N, Tofique S, Kiran T, Pierce M, Chaudhry IB, Husain MO, Memon R, Waqas A, Gire N, Edwards S, Bassitt P, Shakoor S, Zaddeh ZF, Arshad U, Colucci E, Mughal F, Shahid S, Panagioti M, Nizami AT, Jafri F, Naeem F, Emsley R, Ansari MA, Sultan S, Aggarwal S, Williams C, Chaudhry N. Effectiveness of YCMAP (youth culturally adapted manual assisted problem solving) intervention in adolescents after self-harm in Pakistan: multicentre, randomised controlled trial. BMJ. 2025 Sep 12;390:e083272. doi: 10.1136/bmj-2024-083272. PMID 40940081
- [Derived] Husain N, Tofique S, Chaudhry IB, Kiran T, Taylor P, Williams C, Memon R, Aggarwal S, Alvi MH, Ananiadou S, Ansari MA, Aseem S, Beck A, Alam S, Colucci E, Davidson K, Edwards S, Emsley R, Green J, Gumber A, Hawton K, Jafri F, Khaliq A, Mason T, Mcreath A, Minhas A, Naeem F, Naqvi HA, Noureen A, Panagioti M, Patel A, Poppleton A, Shiri T, Simic M, Sultan S, Nizami AT, Zadeh Z, Zafar SN, Chaudhry N. Youth Culturally adapted Manual Assisted Problem Solving Training (YCMAP) in Pakistani adolescent with a history of self-harm: protocol for multicentre clinical and cost-effectiveness randomised controlled trial. BMJ Open. 2022 May 13;12(5):e056301. doi: 10.1136/bmjopen-2021-056301. PMID 35568489
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Interventions for self-harm in children and adolescents. Cochrane Database Syst Rev. 2021 Mar 7;3(3):CD013667. doi: 10.1002/14651858.CD013667.pub2. PMID 33677832
- See also: Pakistan Institute of Living and Learning — http://pill.org.pk